CLINICAL TRIAL: NCT04715542
Title: Subcutaneous Stibium Metallicum Praeparatum 6x Versus Placebo in the PRevention Of PaclitaxEL-induced Peripheral NeurOTOXicity: the PROPEL NO TOX Randomized Controlled Trial
Brief Title: Stibium Metallicum Praeparatum 6x Versus Placebo in the Prevention of Paclitaxel-induced Peripheral Neurotoxicity
Acronym: PROPEL NO TOX
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Hospital of Thun (Unknown); Tumor- und BrustZentrum Ostschweiz (Unknown); Gesundheitszentrum Fricktal AG (Unknown); Kantonsspital Winterthur KSW (Other); Kantonsspital Graubünden (Other); Kantonsspital Aarau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12012021
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Intervention Model Description: Randomized-controlled, double-blind, multicentric superiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stibium metallicum praeparatum 6x (Experimental): Patients are treated with Stibium metallicum praeparatum 6x (subcutaneus injection), which is authorized in Switzerland and is listed by Swissmedic as an authorized anthroposophic medicinal product.
  Interventions: Drug: Stibium metallicum praeparatum 6x
- Saline subcutaneous injection (Placebo Comparator): Placebo (a saline subcutaneous injection) is chosen as comparator to the treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Stibium metallicum praeparatum 6x — Stibium metallicum praeparatum 6x will be administered with subcutaneous injections 3 times a week at 1 ampoule at 1 mL during the chemotherapy and shall be continued during 6 weeks after the end of chemotherapy . The first injection will be administered on the day of the first dose of chemotherapy, before the injection of the first dose of chemotherapy.
  Arms: Stibium metallicum praeparatum 6x
Drug: Placebo — Placebo will be administered with subcutaneous injections 3 times a week at 1 ampoule at 1 mL during the chemotherapy and shall be continued during 6 weeks after the end of chemotherapy . The first injection will be administered on the day of the first dose of chemotherapy, before the injection of the first dose of chemotherapy.
  Arms: Saline subcutaneous injection

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) is one of the most limiting side effects of chemotherapy and often leads to adaptations in the protocol of the chemotherapy including dose reduction or even discontinuation of treatment. In general, the symptoms of CIPN are sensory, often distributed in a "stocking and glove" manner, and include pain, tingling, and numbness. CIPN has a marked negative influence on quality of life of patients and their families. It may result in serious limitations in daily functioning and affect the enjoyment, social relationships, and ability to perform work. Current management of CIPN (i.e. prevention and treatment) includes dose reduction or delay of chemotherapy cycles and treatment discontinuation. Unfortunately, this reduces the chance of an effective cancer treatment. Current guidelines of the American Society of Clinical Oncology (ASCO) on the Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy do not conclusively recommend any agent for the prevention of CIPN. Due to the scarcity of drugs that are effective for preventing and treating CIPN, the distress of patients who suffer from CIPN, and the major societal and economic costs, new approaches and effective treatment strategies are required.

The proposed trial is a parallel, double blind, placebo controlled, randomised, phase III superiority trial, aiming to determine whether treatment with SMP prevents incidence of or reduces the severity symptoms of paclitaxel-induced peripheral neuropathy, as compared to placebo.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most limiting side effects of chemotherapy and often leads to adaptations in the administration of the chemotherapy, including dose reduction or even discontinuation of treatment. In general, the symptoms of CIPN are sensory, often occuring in a "stocking and glove" manner, and most commonly including tingling, numbness, and dysaesthesia. In addition, patients treated with agents inducing CIPN, such as taxanes or platinum compounds, also may experience motor symptoms, which often present as distal or general weakness, and autonomic nervous system dysfunction (e.g. constipation or diarrhea, abnormalities of sweating, and lightheadedness and/or dizziness with positional changes). Furthermore, patients with chronic symptoms report having unsteady gait, putting them at higher risk of falling. CIPN has a largest impact on quality of life and is associated with the development of psychological distress. Cancer survivors' report long-term peripheral neuropathy symptoms with impact on symptom burden, functional status, and quality of life. Because of the growing prevalence of cancer and of cancer survivors, the lack of adequate treatment or preventive strategies against CIPN, as well as the major societal and economic costs, CIPN is becoming a major issue.

According to the National Comprehensive Cancer Network (NCCN) task force report, the overall incidence of CIPN ranges from 57 up to 83% of patients treated with paclitaxel. The incidence and prevalence of CIPN vary among neurotoxic agents, dosing regimens (intensity and cumulative dosing), regimen selection (e.g. combination taxanes and platinum compounds), as well as in presence of preexisting neuropathy, comorbidities and genetic susceptibility. The analysis of the Japanese Adverse Drug Event Report database showed that more than 50% of CIPN associated with taxanes and platinum compounds occurred within four weeks.

After completion of chemotherapy, the prevalence of CIPN for neurotoxic chemotherapy overall one month after finishing chemotherapy is 68%, dropping to 60% at 3 months and 30% at 6 months or more. Severe symptoms are likely to persist longer. In patients treated with taxanes, nearly half of patients have symptoms 6 to 9 months after completing chemotherapy, and many require years to recover, if they recover at all. In early-stage breast cancer patients treated with paclitaxel, persistent numbness one year after treatment with paclitaxel were reported in approximately 67% to 80% of early-stage breast cancer patients. Two years after the end of therapy, 34.4% of breast cancer patients treated with paclitaxel reported neuropathy symptoms, with 18.0% reporting more severe symptoms. Another study showed that two or more years after diagnosis, 44% of breast cancer survivors treated with paclitaxel reported long-term neuropathy symptoms.

Current standard of care Current management of CIPN (i.e. prevention and treatment) includes dose reduction, delay of chemotherapy cycles, or treatment discontinuation. This reduces the chance of an effective cancer treatment.

The 2014, 2020, and 2021 American Society of Clinical Oncology (ASCO) Guidelines on the Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy did not recommend any agent for the prevention of CIPN, and have cautiously recommended treatment of existing CIPN with duloxetine. Preliminary evidence suggests a potential benefit from non-pharmacological treatments in the prevention and/or treatment of chronic neuropathy including exercise, acupuncture, cryotherapy, compression therapy, and scrambler therapy. Larger sample-sized definitive studies are needed to confirm efficacy and clarify risks of these interventions.

Risk factors for CIPN Cumulative dose is a strong risk factor for the development of CIPN. Other risk factors include dose per cycle, treatment schedule (number of injections), duration of infusion, prior or concomitant chemotherapy with neurotoxic agents (i.e. vinca alkaloids, taxanes, platinum compounds, epothilones including ixabepilone, bortezomib, thalidomide, arsenice trioxides), development and severity of acute neuropathy syndrome or acute pain syndrome within 1 to 4 days following the neurotoxic agent infusion, comorbid health conditions associated with an increased risk of neuropathy (i.e. diabetes mellitus, excess alcohol, HIV, smoking, decreased creatinine clearance, folate/vitamin B12 deficiency), pre-existing peripheral neuropathy, older age, and higher body mass index. Other clinical risk factors such as sedentary behavior, insomnia, fatigue, anxiety, and depression have been shown to increase CIPN prevalence. Genetic factors may also be associated with risk of developing CIPN.

Research question Due to the scarcity of drugs that are effective for preventing and treating CIPN, the distress of patients who suffer from CIPN, and the major societal and economic costs, new approaches and effective treatment strategies are required. This study investigates the efficacy and tolerance of Stibium metallicum praeparatum 6x (Weleda), also known as Antimon, to prevent paclitaxel-induced peripheral neuropathy as reported by patients. As secondary outcomes, the influence on quality of life, pain, anxiety, depression, patient's distress, sleep disorder, falls, as well as on chemotherapy treatment adherence and dose of chemotherapy delivered is assessed.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18
* Individuals with early breast cancer, stage I to IIIC, who are about to receive a paclitaxel-based neo-adjuvant or adjuvant chemotherapy, with a planned dosing regimen of 80 mg of paclitaxel per square meter of body surface by intravenous infusion weekly for 12 doses.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Ability to provide informed consent as documented by signature
* Ability to read, write, and speak German

Exclusion Criteria:

* Patients with pre-existing neuropathy
* Prior chemotherapy with taxanes or other neurotoxic agents
* Concomitant medications that are known to cause neuropathy
* Pregnancy or lactation
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Patients with psychiatric, addictive or any disorder that prevents the patient from adhering to the protocol requirements, in the opinion of the investigator
* Lactose intolerance or glucose-galactose-malabsorption, as well as any other contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in neuropathy severity | Week 18
  Measured by the neurotoxicity subscale (NTX-subscale) of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX)

SECONDARY OUTCOMES:
Reduction of occurrence (incidence) of paclitaxel- or nab-paclitaxel-induced peripheral neuropathy | Baseline, Week 3, Week 6, Week 9, Week 12, Week 18; Follow up: Weeks 24, 36, 48, 60
  Measured as per the statistical analysis protocol
Benefit of study medication on Quality of life | Baseline, Week 3, Week 6, Week 9, Week 12, Week 18; Follow up: Weeks 24, 36, 48, 60
  Measured using the 27-item questionnaire FACT-G
Benefit of study medication on pain | Baseline, Week 3, Week 6, Week 9, Week 12, Week 18; Follow up: Weeks 24, 36, 48, 60
  Measured with the Brief Pain Inventory (BPI).
Benefit of study medication on depression | Baseline, Week 12, Follow up: Weeks 24, 36, 48, 60
  Measured with the Patient Health Questionnaire (PHQ-9)
Benefit of study medication on anxiety | Baseline, Week 12, Follow up: Weeks 24, 36, 48, 60
  Measured with the General Anxiety Disorder-7 (GAD-7)
Benefit of study medication on psychological distress | Baseline, Week 3, Week 6, Week 9, Week 12, Week 18; Follow up: Weeks 24, 36, 48, 60
  Measured with the NCCN Distress Thermometer (0-10)
Chemotherapy adherence | Baseline, Week 3, Week 6, Week 9, Week 12, Week 18
  Chemotherapy adherence of patients will be recorded by the study nurse

OTHER OUTCOMES:
Adherence to study medication | Baseline, Week 3, Week 6, Week 9, Week 12, Week 18
  Measured by the total number of unused study drugs returned by the patient
Severe adverse events | Baseline, Week 3, Week 6, Week 9, Week 12
  Any (serious) adverse event (AE) will be recorded, including time of onset, duration, resolution, action to be taken, assessment of intensity and relationship with study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wolf, Prof. Dr., Study Director — University of Bern; Manuela Rabaglio, Dr. med., Principal Investigator — University of Bern; Christoph Ackermann, Dr. med., Principal Investigator — Hospital Thun

IPD SHARING:
Plan to Share IPD: No
IPD will never be available to other researchers who are not part of the core research group. Unblinding is explicitly not foreseen for this study. Maintaining blinding until all participants complete the study protocol, the data base is locked and analysis is completed, will help retain trial integrity of this double-blinded study.